CLINICAL TRIAL: NCT02381171
Title: Transcranial Magnetic Stimulation and/or Neurofunctional Electrical Acupuncture in the Rehabilitation of Patients With Myofascial Chronic Pain
Brief Title: Transcranial Magnetic Stimulation and/or Neurofunctional Electrical Acupuncture in Myofascial Chronic Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Spaulding Rehabilitation Hospital (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Wolnei Caumo, The investigation of the effect of transcranial magnetic stimulation and / or Neurofunctional Electrical Acupuncture in the rehabilitation of patients with myofascial chronic pain, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HCPA-TMS
Record Dates: First submitted 2014-03-21; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Myofascial Pain Syndromes
Keywords: myofacial pain; neuromodulation; repetitive transcranial magnetic stimulation; electroacupuncture
MeSH Terms: conditions — Myofascial Pain Syndromes; Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Both Sham rTMS and Neuroacupuncture (Sham Comparator): Subjects will be randomized to receive 10 sessions of both sham treatments. Stimulation will be given on consecutive days (Monday- Friday) for 2 weeks: rTMSat 10hHz (1600pulses) over the primary motor cortex area and neurofunctional electrical acupuncture without current connection over peripheral region.
  Interventions: Device: Sham rTMS; Device: Sham Neuroacupuncture
- Active rTMS and sham Neuroacupuncture (Sham Comparator): Subjects will be randomized to receive 10 sessions of active rTMS and sham neurofunctional electrical acupuncture treatments. Stimulation will be given on consecutive days (Monday- Friday) for 2 weeks: rTMS at 10Hz (1600 pulses) over the primary motor cortex area and neurofunctional electrical acupuncture without current connection over peripheral region.
  Interventions: Device: Active rTMS; Device: Sham Neuroacupuncture
- Sham rTMS and Active Neuroacupuncture (Sham Comparator): Subjects will be randomized to receive 10 sessions of sham rTMS and active Neurofunctional Electrical Acupuncture. Stimulation will be given on consecutive days (Monday- Friday) for 2 weeks: rTMS placebo coil over the primary motor cortex area and neurofunctional electrical acupuncture at 1Hz, continuous, 10mA current for 20 minutes over peripheral region.
  Interventions: Device: Sham rTMS; Device: Active Neuroacupuncture
- Both Active rTMS and Neuroacupuncture (Active Comparator): Experimental Subjects will be randomized to receive 10 sessions of both active treatments. Stimulation will be given on consecutive days (Monday- Friday) for 2 weeks: rTMS at 10 Hz (1600 pulses) over the primary motor cortex area and neurofunctional electrical acupuncture at 1Hz, continuous, 10mA current for 20 minutes over peripheral region.
  Interventions: Device: Active rTMS; Device: Active Neuroacupuncture

INTERVENTIONS:
Device: Active rTMS — Repetitive Transcranial Magnetic Stimulation (rTMS) 10Hz (1600 pulses)
  Arms: Active rTMS and sham Neuroacupuncture; Both Active rTMS and Neuroacupuncture
Device: Sham rTMS — Repetitive Transcranial Magnetic Stimulation (rTMS) with Placebo coil
  Arms: Both Sham rTMS and Neuroacupuncture; Sham rTMS and Active Neuroacupuncture
Device: Active Neuroacupuncture — Neurofunctional electrical acupuncture 1Hz, continuous, 10mA current for 20 minutes.
  Other Names: Electrical Deep Intramuscular Stimulation
  Arms: Both Active rTMS and Neuroacupuncture; Sham rTMS and Active Neuroacupuncture
Device: Sham Neuroacupuncture — Neurofunctional electrical acupuncture without needles
  Other Names: Sham Electrical Deep Intramuscular Stimulation
  Arms: Active rTMS and sham Neuroacupuncture; Both Sham rTMS and Neuroacupuncture

SUMMARY:
To evaluate the hypothesis: the effects of repetitive transcranial magnetic (rTMS) stimulation and/or peripheral stimulation (neurofunctional electrical acupuncture) treatments are more effective in pain relief than placebo-sham in patients with myofascial chronic pain.

DETAILED DESCRIPTION:
This project is a multidisciplinary study, with available technology, which aims are to provide more data to consolidate the techniques of central and peripheral neuromodulation in the treatment of myofascial pain with a component in the craniofacial complex . This is a randomized, double-dummy, factorial, blind, parallel, placebo - sham controlled clinical trial. The issues investigated in this study include important public health problem because chronic musculoskeletal pain affects 30 % of the world population , according to WHO. Around 75-80 % of people seeking health care for pain and that 40% of adults suffer from some type of chronic pain. According to the severity of the problem , the International Association for the Study of Pain has defined the year 2010 as the International Year Against Musculoskeletal Pain, facing the increasing prevalence and the limited impact of the classical therapeutic interventions ( ~ 30 % ). Possibly, part of this poor response is due to the limitation of pathophysiological knowledge, few resources in diagnostic methods and the consequent implementation of measures that do not reach the main routes of this disease process. It is important to mention that epidemiological studies have greatly contributed to improve the understanding of the process of these musculoskeletal diseases, but increase few knowledge about the understanding of the pathophysiology, diagnostic and therapeutic developments. It is important to highlight that evidence has shown strong association of musculoskeletal pathologies conditions and chronic stress. This relationship is cascading and permeated by manifestations suggest that the neuro-immune-endocrine axis, such as poor sleep quality, anxiety symptoms, depressive symptoms, increased susceptibility to infections and manifestations of neuro-vegetative dysfunctions. Thus, this project will examine whether the hypothesis that the application of central and peripheral neuromodulatory therapies can have a positive impact on possible systems implicated in the pathophysiological course of musculoskeletal disorders in the craniofacial complex, and evaluate clinical outcomes characterizing the process of rehabilitation of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent to participate in the study ;
* 18 to 70 years old;
* Myofascial pain in the cranial- cervical- mandibular complex, with duration more than 3 months;
* In the last week, score higher or equal to 3cm (0 cm = 'no pain' and 10cm ='worst possible pain') on the VAS for pain perception at the baseline in the most part of seven days before;
* Refractoriness to drugs for pain relieve - such as tricyclic antidepressants, antiepileptic drugs and/or narcotics (pain resistant to at least 2 of these drugs supplied in adequate dosages for six months).

Exclusion Criteria:

* Inflammatory chronic disease;
* Neurological deficits;
* History of substance abuse;
* Neuropsychiatric co-morbidity;
* Systemic diseases not well balance;
* Habitual use of anti-inflammatory steroids;
* Implanted devices for pain control, such as vagal or deep brain stimulators;
* Contraindications to rTMS: metal in the head, implanted brain medical devices, previous convulsion or epilepsy, serious cranial trauma, audition problem, cochlear implant, neurostimulador implantable, spinal cord surgery, bypass valve ventriculoperitoneal peritonenal,cardiac pacemaker or other metal in the body;
* Pregnancy;
* Prior experience with acupuncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain severity | up to three months after the end of treatment
  The intensity of pain was measured by a 10-cm VAS. VAS scores ranged from no pain (zero) to the worst possible pain (10cm).

SECONDARY OUTCOMES:
Peripheral Biochemical Markers | The difference in the baseline, after one week of treatment and the end of the treatment (2 weeks after starting the treatment).
  Different peripheral biochemical: BDNF, TNF, S100 beta, interleukins, LDH, oxidative stress, catecolamines serum levels; 6-sulphatoxymelatonin urinary; salivary cortisol.
Parameters of motor cortex excitability | The variation between the baseline and the end of treatment (2 weeks after starting the treatment).
  Parameters of cortical excitability: motor threshold, motor-evoked potential, intracortical inhibition and facilitation, cortical silent period using transcranial magnetic stimulation technique.
Quality of Life | Baseline (before the treatment) and after the treatment (after last session of treatment and follow-up of two weeks, one month and three months after the end of treatment )
  Using Quality of life questionnaire (WHOQOL-bref) with 26 questions.
Functional Capacity | Baseline (before the treatment) and after the treatment (after last session of treatment and follow-up of two weeks, one month and three months after the end of treatment ).
  Using The Brazilian Portuguese version of the Profile of Chronic Pain.
Pain threshold | The variation between the baseline and the end of treatment (2 weeks after starting the treatment).
  Pain threshold assessed by algometer (pain pressure threshold) and quantitative sensory

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Botelho L, Angoleri L, Zortea M, Deitos A, Brietzke A, Torres ILS, Fregni F, Caumo W. Insights About the Neuroplasticity State on the Effect of Intramuscular Electrical Stimulation in Pain and Disability Associated With Chronic Myofascial Pain Syndrome (MPS): A Double-Blind, Randomized, Sham-Controlled Trial. Front Hum Neurosci. 2018 Oct 16;12:388. doi: 10.3389/fnhum.2018.00388. eCollection 2018. PMID 30459575
- [Derived] Medeiros LF, Caumo W, Dussan-Sarria J, Deitos A, Brietzke A, Laste G, Campos-Carraro C, de Souza A, Scarabelot VL, Cioato SG, Vercelino R, de Castro AL, Araujo AS, Bello-Klein A, Fregni F, Torres IL. Effect of Deep Intramuscular Stimulation and Transcranial Magnetic Stimulation on Neurophysiological Biomarkers in Chronic Myofascial Pain Syndrome. Pain Med. 2016 Jan;17(1):122-35. doi: 10.1111/pme.12919. PMID 26408420